CLINICAL TRIAL: NCT03255720
Title: Application of Diffusion Tensor Imaging in Alzheimer's Disease:Quantification of White Matter Micro-structural Changes
Brief Title: Application of Diffusion Tensor Imaging in Alzheimer's Disease :Quantification of White Matter Micro-structural Changes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, shereen magdy, principal investigator, Assiut University
Other Study IDs: diffusion tensor imaging
Record Dates: First submitted 2017-08-15; First posted 2017-08-21 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Alzheimer Dementia
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 20 patients with Alzheimer disease: The study will be performed at the Radiodiagnosis department of assiut university hospital.
  Selection of 20 patients clinically and laboratory diagnosed as Alzheimer disease and another 20 people matched healthy controls who have no complaints of cognitive problems.
- 20 people matched healthy controls: health control people who have no complaints of cognitive problems.

SUMMARY:
Diffusion Tensor imaging of white matter degeneration in Alzheimer disease

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common cause of dementia in the elderly, accountings for 60-70% of all demented cases. It is a neuro-pathological diagnosis determined by presence of neurofibrillary tangles and senile plaques in the brain of patients with dementia. The disease frequently starts with memory impairment, but is invariably followed by a progressive global cognitive impairment. The major risk factor for Alzheimer disease is age, with prevalence doubling every 5 years after the age of 65.

Diagnosis of Alzheimer's typically involves physical and neurological exams, as medical history and mental status evaluation, laboratory investigations and it involves brain imaging (such as MRI) which could identify other causes of problems such as stroke, tumor or head trauma. By physical and neurological examination, Alzheimer's disease characterized by gradual onset and progressive decline in cognition with sparring of motor and sensory function until later stages; the average course of Alzheimer's disease is approximately a decade, with a range of 3 to 20 years duration from diagnosis to death .Memory impairment is present in the earliest stages of the disease; patients have difficulty learning new information and retaining it for more than few minutes. As the disease advances, the ability to learn increasingly compromised, more distant memories are lost. Other cognitive loses include aphasia, apraxia, disorientation and impaired judgment. Cognitive impairment affects daily life; patients have difficulty planning meals, managing finances or medication, using telephone, driving. Many capacities may remain intact until later stages including performance of self-care activities of daily living as eating, bathing. Patients evidence personality alteration, irritability, anxiety, depression. Delusion, hallucination and aggression. Laboratory Evaluation includes Biochemical markers as measurement of Cerebrospinal fluid including Tau protein, amyloid beta peptides or neural thread protein and measurement of urinary biomarkers including neural thread protein. Also testing including Apo lipoprotein E epsilon 4 allele presenilin genes, amyloid precursor gene or TREM2. Diffusion tensor imaging (DTI) is an imaging technology based on magnetic resonance diffusion weighted imaging, which can make quantitative analysis of anisotropy of water molecules in different directions, so as to observe the microstructure of tissues non-invasively. So Diffusion tensor imaging can provide information of fiber orientation, the injury of fiber, and membrane permeability which cannot be obtained from conventional MRI. Diffusion tensor imaging enables mapping of White matter microstructure changes in development, aging and neurological disorders, From the tensor, it's possible to derive the mean diffusivity (DM) and the fractional anisotropy (FA) which is the most robust measures of anisotropy which measure the degree of deviation from isotropic diffusion. ). More recently, an additional DT-MRI derived index has been proposed .This index measures the degree of similarity of orientation of neighboring voxels and its named inter-voxel coherence (C).

So Diffusion tensor imaging has therefore become a powerful technique in the study of neurodegenerative diseases in recent years.

ELIGIBILITY:
Inclusion Criteria:

1. cognitive complaints with interference in complex occupational and social activities.
2. changes in cognition reported by the patient ,informant or clinician.
3. absence of profound sub-cortical ischemic changes.

Exclusion Criteria:

1. state of delirium
2. stroke event within 2 weeks
3. appearance of cortical and /cortico-subcortical non -lacunar territorial infarcts and watershed infarcts ,hemorrhage ,signs of normal pressure hydrocephalus ,and specific causes of white matter lesions (e.g. multiple sclerosis, sarcoidosis, brain irradiation)
4. derangements in serology tests contributing to cognitive impairment (e.g. abnormal levels of free T4 or rapid plasma reagin.
5. severe hearing or visual impairment.
6. cases of severe dementia.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: old aged people over 60 years
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-09-29 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
the extent of tissue damage of several brain white matter regions in patients with Alzheimer's disease. | 4 years
  provide a complete picture of the distribution of microstructural white matter damage in Alzheimer's disease

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT03255720/Prot_000.pdf